CLINICAL TRIAL: NCT02029781
Title: APPLE Study (APPendicitis and Laparoscopic Evaluation) Study; Multicenter Prospective Validation of the Laparoscopic APPendicitis (LAPP) Score
Brief Title: The Laparoscopic Appendicitis Score; a Multicenter Validation Study
Acronym: APPLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delayed/poor inclusion rate.
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Groningen (Other)
Responsible Party: Principal Investigator, JW Haveman, MD, PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Apple study 2013
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Appendicitis
Keywords: Appendicitis; Laparoscopy; Appendectomy; Negative appendectomy; Morbidity
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LAPP score (Other): Use of the LAPP score during a diagnostic laparoscopy.
  Interventions: Procedure: LAPP score

INTERVENTIONS:
Procedure: LAPP score — Use of the LAPP score during a diagnostic laparoscopy.

SUMMARY:
SUMMARY

Rationale: A diagnostic laparoscopy is a frequently used method to confirm the diagnosis appendicitis. However until recently evidence-based laparoscopic criteria for determining appendicitis were not defined. If there is any doubt about the presence of appendicitis the appendix is usually removed. In a single centre prospective pilot study on 134 patients the investigators were able to define the Laparoscopic APPendicitis (LAPP) score. In the current study the investigators will validate the LAPP score in order to decrease the negative appendectomy rate by 50%. Eventually the score should lead to a decrease in morbidity.

Objective: To decrease the negative appendectomy rate by 50%.

Study design: A multicenter prospective validation study

Study population: All patients, ≥18 years, operated with a diagnostic laparoscopy for the clinical suspicion appendicitis. Sample size calculation, performed by a statistician/ epidemiologist of the Trial Coordination Centre, showed the need to analyse 778 patients.

Intervention (if applicable): Patients operated on appendicitis in 2008 and 2009 (n=843), were retrospectively analysed for negative appendectomies. This cohort will serve as the control group. In this control group no intervention was given, as the LAPP score was not yet defined.

In the 778 prospective analysed patients, the LAPP score will be used during a diagnostic laparoscopy. With the LAPP score the investigators intend to halve the number of negative appendectomies.

Main study parameters/endpoints: A decrease in the negative appendectomy rate from 9% to 5%. This decrease should not lead to an increase in missed appendicitis (occurring within 30 days), defined as requiring a surgical re-intervention or as an appendicitis or appendicular infiltrate on an ultrasound or CT-scan.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risk of implementation of the LAPP score is minimal. In theory, the use of the LAPP score might lead to an increase risk in missed appendicitis. This might lead to an increase in morbidity.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE

   During the last decade, a laparoscopic approach for a suspicion of appendicitis has become more common in surgical practice. In case the appendix looks normal the guideline of the Dutch Society of Surgeons advices not to remove it. [1] The morbidity of a negative appendectomy is approximately 6% and it also leads to additional costs. [2] However, until recently no criteria on how to assess the appendix during a laparoscopy has been published. In a recently performed pilot study the investigators defined the Laparoscopic APPendectomy (LAPP) score. [3] The LAPP score is an easy applicable score that can be used during a diagnostic laparoscopy to evaluate the appendix on the presence or absence of 5 laparoscopic criteria on appendicitis. In our prospective cohort, use of the LAPP score would have led to a positive predictive value of 99% and a negative predictive value of 100%.

   The goal of the current study is to validate the LAPP score in a prospective multicenter validation study. Our hypothesis is that the application of the LAPP score leads to a reduction of 50% of negative appendectomies compared with a retrospective cohort in the same centers. The investigators have chosen to compare the negative appendectomy rate of this prospective multicenter validation study with a retrospective control group. The control group consists of 843 patients operated in 5 centers in 2008 and 2009 with a negative appendectomy rate of 9%.

   The most ideal design would be a clustered center randomized trial. In such a case half of the hospitals will be asked to use the LAPP score and the other half should assess the appendix the conventional way. The investigators feel that it is not feasible, as they already presented the LAPP score at the national congress for surgeons. In addition, after publication of the results of the LAPP study surgeons might already start to use the LAPP score or at least will evaluate the appendix differently than before. [3]
2. OBJECTIVES

   Primary Objective: To reduce the negative appendectomy rate with 50% compared with the retrospective control group.

   Secondary Objective(s):
   * The percentage of missed appendicitis should not exceed 1%.
   * Analyse sensitivity rate.
   * Cost from used materials during the operation.
   * Cost form the histology review by the pathologist of a removed appendix
3. STUDY DESIGN

   Prospective cohort design, multicenter prospective validation study in 778 patients suspected for appendicitis with an indication for diagnostic laparoscopy. The investigators expect to fulfill the inclusion within one and half year.

   This cohort will be compared with a multicenter historical cohort. Each center will be its own control group.
4. STUDY POPULATION

   Population (base) All patients operated for the suspicion of acute appendicitis. The preoperative work-up is not standardized for this study; therefore the investigators stick to the protocol of each hospital. The clinical decision to operate the patient will be made by the surgeon on call. Only patients that will undergo a (diagnostic) laparoscopy can be included in this study.

   A total of 778 patients must be included. The investigators intend to fulfill inclusion within one and a half year. This duration is based on prevalence of appendicitis in the Netherlands. Annually, 16.000 appendectomies are performed, in combination with eight participating centers, the investigators think this is a feasible period.

   Sample size calculation The sample size calculation was performed according to the methods by William D. Dupont and Walton D. Plummer (PS Power and Sample Size Calculations). For the sample size calculation the investigators performed a retrospective cohort analysis in 2008 and 2009 in 5 hospitals in the Netherlands (Wilhelmina Ziekenhuis Assen, Nij Smellinghe Ziekenhuis Drachten, Universitair Medisch Centrum Groningen, Medisch Centrum Leeuwarden and Martini Ziekenhuis Groningen). During this period 843 patients were operated for the suspicion of acute appendicitis with a diagnostic laparoscopy, 9% of the removed appendices turned out to be normal (appendix sana). In order to half the negative appendectomy rate with a power of 0.8 and an alpha of 0.05, 544 patients in the prospective group are needed. Our previous prospective analysis (the LAPP study) and the retrospective data showed that approximately 15% of the included patients will have another diagnosis (Crohn's disease, ruptured ovarian cyst etc.), additionally the investigators expect another 15% of exclusions because for example no clear laparoscopic view of the appendix (figure 1). Therefore the investigators need 778 patients in our multicenter prospective validation study.

   Important to mention, in the sample size calculation they did not take sensitivity rate into account, as they expect the sensitivity will be around 100%. However, the investigators will calculate this percentage and report is in the results section.
5. TREATMENT OF SUBJECTS

   5.1 Investigational product/treatment Use of the LAPP score. The LAPP score consists of 5 questions concerning criteria of appendicitis, if 1 or more of these questions are answered with 'yes' the appendix should be removed, if all questions are answered with 'no' the appendix should not be removed.

   The five questions are:
   * Is there perforation and/or necrosis of the appendix;
   * Is the appendix thickened;
   * Is the mesentery of the appendix thickened;
   * Is there presence of injected vessels on the serosa of the appendix;
   * Are there any adhesions around the appendix.

   5.2 Use of co-intervention (if applicable) Not applicable

   5.3 Escape medication (if applicable) Not applicable.
6. INVESTIGATIONAL PRODUCT

   Not applicable, as this study concerns no research with medicinal products.
7. NON-INVESTIGATIONAL PRODUCT

   Not applicable
8. METHODS

   8.1 Study parameters/endpoints 8.1.1 Main study parameter/endpoint The main endpoint of the study is to reduce the negative appendectomy rate with 50%. The gold standard is the histological examination by the pathologist. The pathologist considers the appendix as inflamed when at least (local) ulceration with infiltration of polymorphonuclear neutrophils into the mucosa and submucosa (endo-appendicitis) is present, either or not in combination with transmural inflammation, necrosis, perforation and peri-appendicular inflammation. In case of inflammation without mucosal ulceration was found, the contralateral part of the appendix and more transverse slices were examined. [4] An appendix is considered as normal when no signs of inflammation are found and when no other abnormality is found like more rare entities as carcinoid, adenocarcinoma of the appendix or a parasite infection.

   8.1.2 Secondary study parameters/endpoints (if applicable)
   * The percentage of missed appendicitis; this should not exceed 1%. In theory the LAPP score might lead to an increase in missed appendicitis. This might happen when a patient has an early or mild appendicitis without any of the 5 laparoscopic criteria for appendicitis. The investigators have defined 'missed appendicitis' as a confirmed appendicitis or appendicular infiltrate on a CT-scan or during a re-operation (within 3 months).
   * Cost from used material during the operation.
   * Cost form the histology review by the pathologist of a removed appendix.

   8.1.3 Other study parameters (if applicable) Not applicable

   8.2 Randomisation, blinding and treatment allocation All included patients will undergo a diagnostic laparoscopy, during this procedure the LAPP score will be used and on the basis of the results the appendix will be removed or not.

   8.3 Study procedures There are no additional procedures the patients will undergo during this study.

   8.4 Withdrawal of individual subjects Subjects can leave the study at any time for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject from the study for urgent medical reasons.

   8.4.1 Specific criteria for withdrawal (if applicable) For whatever reason the patient is free to withdraw from the study. After the patient is asked to participate in the study in the emergency department or on the surgical ward and has signed the informed consent form, he/she will usually have to wait for some time before he/she is operated on. In theatre the LAPP score will be used. Postoperatively the patient can still decide to withdraw from the study, although the decision to remove or not to remove the appendix has already been made. The patient will be prospective followed for 12 months and during this period the patient can still decide to withdraw from the study, then all saved data and forms will be deleted from the database.

   8.5 Replacement of individual subjects after withdrawal There is no need to replace a patient that has withdrawn. In our sample size calculation the investigators anticipated a 40% rate of withdrawal for several reasons.

   8.6 Follow-up of subjects withdrawn from treatment These patients will have the usual follow-up for patients operated on for the suspicion of appendicitis. In most case patients will be seen postoperatively once or twice in the outpatient clinics.

   8.7 Premature termination of the study
   * At 2 different time intervals, when 50 and 75% of the total number of patients are included in the study an interim analysis will be performed. The percentage of missed appendicitis will be evaluated. When the percentage of missed appendicitis exceeds 2%, the study will be terminated.
   * The percentage of missed appendicitis leading to a serious adverse event (like persistent or significant disability or incapacity, life threatening or death) should not exceed 1%. This will be evaluated at any time during the study.
9. SAFETY REPORTING

9.1 Section 10 WMO event In accordance to section 10, subsection 1, of the WMO, the investigator will inform the subjects and the reviewing accredited METC if anything occurs, on the basis of which it appears that the disadvantages of participation may be significantly greater than was foreseen in the research proposal. The study will be suspended pending further review by the accredited METC, except insofar as suspension would jeopardise the subjects' health. The investigator will take care that all subjects are kept informed.

9.2 AEs, SAEs and SUSARs 9.2.1 Adverse events (AEs) See also section 8.7. Serious adverse events caused by a missed appendicitis will be reported immediately when they occur. If a missed appendicitis leads to a prolongation of hospitalization of less than 10 days the investigators will consider this as an adverse event and take no further action unless this exceeds 2% after inclusion of every quartile of patients.

Adverse events like persistent or significant disability or incapacity, life threatening or death will be reported immediately or at least within 7 days to the web portal ToetsingOnline.

Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to [the investigational product / the experimental intervention]. All adverse events reported spontaneously by the subject or observed by the investiga¬tor or his staff will be recorded.

9.2.2 Serious adverse events (SAEs)

A serious adverse event is any untoward medical occurrence or effect that at any dose:

* results in death;
* is life threatening (at the time of the event);
* requires hospitalisation or prolongation of existing inpatients' hospitalisation;
* results in persistent or significant disability or incapacity;
* is a congenital anomaly or birth defect;
* Any other important medical event that may not result in death, be life threatening, or require hospitalization, may be considered a serious adverse experience when, based upon appropriate medical judgement, the event may jeopardize the subject or may require an intervention to prevent one of the outcomes listed above.

The sponsor will report the SAEs through the web portal ToetsingOnline to the accredited METC that approved the protocol, within 15 days after the sponsor has first knowledge of the serious adverse reactions.

SAEs that result in death or are life threatening should be reported expedited. The expedited reporting will occur not later than 7 days after the responsible investigator has first knowledge of the adverse reaction. This is for a preliminary report with another 8 days for completion of the report.

9.2.3 Suspected unexpected serious adverse reactions (SUSARs) Not applicable for this study.

9.3 Annual safety report Not applicable for this study.

9.4 Follow-up of adverse events All AEs will be followed until they have abated, or until a stable situation has been reached. Depending on the event, follow up may require additional tests or medical procedures as indicated, and/or referral to the general physician or a medical specialist.

SAEs need to be reported till end of study within the Netherlands, as defined in the protocol.

9.5 [Independent Data Monitoring Committee (IDMC) / Safety Committee] The following doctors will take place in the Independent Data Monitoring Committee;

* Prof. dr. H.W. Nijman, gynaecologist
* Drs. T.H. van Dijk, pediatric surgeon
* Dr. J. Niesing, statistician

ELIGIBILITY:
Inclusion Criteria:

* Patients operated for the clinical suspicion of acute appendicitis that will undergo a diagnostic laparoscopy.
* Age ≥ 18 years.
* Written informed consent

Exclusion Criteria:

* Diagnostic laparoscopy and planned appendectomy for an appendectomy a froid.
* Primarily chosen for an open appendectomy.
* Not able to give informed consent (for example language barrier or legally incapable).
* Refused informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Negative appendectomy | 3 months postoperatively
  Either a histologically proven normal appendix or in case of no appendectomy a 3 months disease free clinical course.

SECONDARY OUTCOMES:
Missed appendicitis | 3 months
  In case the appendix was not removed and the patients developed appendicitis or an infiltrate or appendicular abscess within 3 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided